CLINICAL TRIAL: NCT05052996
Title: A Phase 2 Randomized, Open-Label, Active-Controlled Study Evaluating the Safety and Efficacy of an Oral Weekly Regimen of Islatravir in Combination With Lenacapavir in Virologically Suppressed People With HIV
Brief Title: Study Evaluating the Safety and Efficacy of Islatravir in Combination With Lenacapavir in Virologically Suppressed People With HIV
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-563-6041
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — lenacapavir; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (ISL+LEN) (Experimental): Participants will receive the following for at least 48 weeks:
  * Day 1 and Day 2: ISL 40 and LEN 600 mg
  * Day 8 and weekly thereafter (ie, every 7 days): ISL 20 mg and LEN 300 mg
  Interventions: Drug: ISL; Drug: LEN
- Cohort 1 (B/F/TAF to ISL+LEN) (Experimental): Participants will receive bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg once daily for at least 48 weeks
  After 48 weeks, participants will switch from B/F/TAF to ISL+LEN
  * ISL 40 and LEN 600 mg on Day 1 and Day 2
  * ISL 20 mg and LEN 300 mg weekly
  Participants who do not switch from B/F/TAF to ISL+LEN at Week 48 will be discontinued from the study.
  Interventions: Drug: ISL; Drug: LEN; Drug: B/F/TAF
- Cohort 2 (ISL+LEN) (Experimental): Participants will receive the following for at least 48 weeks
  * Day 1: LEN oral 600 mg (2 x 300 mg) and ISL 2 mg (2 x 1 mg)
  * Day 2: LEN only oral 600 mg (2 x 300 mg)
  * Day 8 and weekly thereafter (ie, every 7 days): LEN oral 300 mg (1 x 300 mg) and ISL 2 mg
  Interventions: Drug: ISL; Drug: LEN
- Cohort 2 (B/F/TAF to ISL+LEN) (Experimental): Participants will receive B/F/TAF 50/200/25 mg once daily for at least 48 weeks.
  Interventions: Drug: ISL; Drug: LEN; Drug: B/F/TAF
- Extension Phase Cohort 2 of ISL/LEN Fixed Dose Combination (FDC) (Experimental): After 48 Weeks of randomized treatment, all participants will be given an option to participate in an Extension Phase to receive ISL+LEN or ISL/LEN FDC tablet (when available) until ISL/LEN becomes available or until the sponsor elects to discontinue the study, whichever occurs first.
  Participants receiving ISL+LEN during the randomized phase will continue to take ISL + LEN weekly.
  Participants receiving B/F/TAF during the randomized phase will switch to ISL+LEN:
  * Day 1: LEN oral 600 mg (2 x 300 mg) and ISL 2 mg (2 x 1 mg)
  * Day 2: LEN only oral 600 mg (2 x 300 mg)
  * Day 8 and weekly thereafter (ie, every 7 days): LEN oral 300 mg (1 x 300 mg) and ISL 2 mg
  Participants who do not switch from B/F/TAF to ISL+LEN at Week 48 will be discontinued from the study.
  All participants in the extension phase will be transitioned to weekly ISL/LEN FDC (Dose A) tablet when it becomes available.
  Interventions: Drug: ISL/LEN FDC

INTERVENTIONS:
Drug: ISL — Capsules administered orally without regard to food
  Arms: Cohort 1 (B/F/TAF to ISL+LEN); Cohort 1 (ISL+LEN); Cohort 2 (B/F/TAF to ISL+LEN); Cohort 2 (ISL+LEN)
Drug: LEN — Tablets administered orally without regard to food
  Other Names: GS-6207
  Arms: Cohort 1 (B/F/TAF to ISL+LEN); Cohort 1 (ISL+LEN); Cohort 2 (B/F/TAF to ISL+LEN); Cohort 2 (ISL+LEN)
Drug: B/F/TAF — Tablets administered orally without regard to food
  Other Names: Biktarvy®
  Arms: Cohort 1 (B/F/TAF to ISL+LEN); Cohort 2 (B/F/TAF to ISL+LEN)
Drug: ISL/LEN FDC — Tablets administered orally without regard to food
  Arms: Extension Phase Cohort 2 of ISL/LEN Fixed Dose Combination (FDC)

SUMMARY:
The primary objective of this study is to evaluate the efficacy of oral weekly islatravir (ISL) in combination with lenacapavir (LEN) in virologically suppressed people with HIV (PWH) at Week 24.

ELIGIBILITY:
Key Inclusion Criteria:

* Received bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) for ≥ 24 weeks at screening.
* Documented plasma human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL) for ≥ 24 weeks before and at screening.
* Plasma HIV-1 RNA < 50 copies/mL at screening.

Key Exclusion Criteria:

* History of prior virologic failure while receiving treatment for HIV-1.
* Prior use of, or exposure to, islatravir (ISL) or lenacapavir (LEN).
* Active, serious infections requiring parenteral therapy < 30 days before randomization.
* Active or occult hepatitis B virus (HBV) coinfection, defined as hepatitis B core antibody (HBcAb) positive, hepatitis B surface antigen (HBsAg) positive, or HBV deoxyribonucleic acid (DNA) positive as determined by the central laboratory.
* Active hepatitis C virus (HCV) coinfection, defined as detectable HCV RNA.
* Any of the following laboratory values at screening:

  * Creatinine clearance (CLcr) ≤ 30 mL/min according to the Cockcroft-Gault formula
* CD4+ T-cells < 200 cells/mm^3 (Cohort 1); CD4+ T-cells < 350 cells/mm^3 (cohort 2).
* Absolute lymphocyte count < 900 cells/mm^3 (cohort 2).
* Individuals of childbearing potential (as defined in protocol) who have a positive serum pregnancy test at screening or positive urine and serum pregnancy tests at Day 1 prior to study drug administration.
* Individuals who plan to continue breastfeeding during the study.
* Documented historical or screening resistance reports showing nucleoside/nucleotide reverse transcriptase inhibitors (NRTIs) or non-nucleoside/nucleotide reverse transcriptase inhibitors (NNRTIs) resistance mutations in reverse transcriptase, including M184V/I (Cohort 2).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2028-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (44):
- United States (44):
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Ruane Clinical Research Group, Inc, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Hoag Medical Group - Newport Beach, Newport Beach, California
  - BIOS Clinical Research, Palm Springs, California
  - Optimus Medical Group, San Francisco, California
  - Public Health Institute at Denver Health, Denver, Colorado
  - Vivent Health, Denver, Colorado
  - Washington Health Institute, Washington D.C., District of Columbia
  - The George Washington University Medical Faculty Associates Inc., Washington D.C., District of Columbia
  - CAN Community Health Care, Inc., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - JEM Research Institute, Lake Worth, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Emory University Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Metro Infectious Disease Consultants, Decatur, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - John A. Burns School of Medicine, University of Hawaii Clinics at Kaka'ako, Honolulu, Hawaii
  - Howard Brown Health Center, Chicago, Illinois
  - Northstar Healthcare, Chicago, Illinois
  - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - Boston Medical Center, Boston, Massachusetts
  - AccessHealth MA, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Hennepin Healthcare HCMC, New Brighton, Minnesota
  - Southampton Healthcare, Inc., St Louis, Missouri
  - Huntridge Family Clinic, Las Vegas, Nevada
  - ID Care, Hillsborough, New Jersey
  - AXCES Research Group, Santa Fe, New Mexico
  - New York-Presbyterian Queens, Flushing, New York
  - Jacobi Medical Center, The Bronx, New York
  - NC TraCS Institute - CTRC: University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Penn Medicine: Perelman Center for Advanced Medicine at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT Community Health Centers, Philadelphia, Pennsylvania
  - Central Texas Clinical Research, LLC, Austin, Texas
  - AIDS Arms Inc, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - The Crofoot Research Center, INC, Houston, Texas
  - Peter Shalit, M.D., Seattle, Washington
  - MultiCare Rockwood Main Clinic, Spokane, Washington
  - Community Health Care, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colson AE, Crofoot GE, Ruane PJ, Ramgopal MN, Dretler AW, Nahass RG, Sinclair GI, Berhe M, Roberts A, Applin S, Brinson C, Jayaweera D, Workowski KA, Shihadeh F, Liu SY, Klopfer S, Llamoso C, Madera S, Dvory-Sobol H, Rhee MS, Rhee EG, Baeten JM, Eron JJ. Once-Weekly Oral Islatravir Plus Lenacapavir Versus Daily Oral Bictegravir, Emtricitabine, and Tenofovir Alafenamide in Persons With HIV-1 : A Phase 2 Randomized Study. Ann Intern Med. 2025 Dec 23. doi: 10.7326/ANNALS-25-01939. Online ahead of print. PMID 41429026
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-563-6041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. This is the primary results analysis including data up to Week 48 for the outcome measures. As Cohort 1 never reached Week 48, so, the data for some outcome measures for applicable timepoints up to Week 48 were reported for Cohort 2 only.
Pre-assignment Details: 322 participants were screened.
Groups:
- Cohort 1- Group 1 (ISL+LEN): Participants received islatravir (ISL) 40 mg and lenacapavir (LEN) 600 mg orally on Days 1 and 2 and ISL 20 mg and LEN 300 mg orally weekly thereafter from Day 8. They were to take treatment up to at least Week 48, however, all participants were off study treatment prior to Week 12 in the study.
- Cohort 1- Group 2 (B/F/TAF to ISL+LEN): Participants received bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg, orally, once daily. They were to take treatment up to Week 48, however, all participants were off study treatment prior to Week 12 in the study.
- Cohort 2- Group 1 (ISL+LEN): Participants received ISL 2 mg and LEN 600 mg orally on Day 1 and 2 and ISL 2 mg and LEN 300 mg orally weekly thereafter from Day 8 for at least 48 weeks.
- Cohort2- Group 2 (B/F/TAF to ISL+LEN): Participants received bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg once daily orally for at least 48 weeks. After 48 weeks, participants will switch from B/F/TAF to ISL+LEN and received ISL 2 mg and LEN 600 mg orally on Day 1 and Day 2, LEN 600 mg orally only on Day 2 and ISL 2 mg and LEN 300 mg orally weekly thereafter from Day 8 for at least 48 weeks.
Period: Overall Study
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Started | 24 | 12 | 53 | 53
Completed | 0 | 0 | 2 | 4
Not Completed | 24 | 12 | 51 | 49
Not completed — Still on study | 0 | 0 | 47 | 44
Not completed — Cohort terminated by sponsor | 21 | 12 | 0 | 0
Not completed — Withdrew consent | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Randomized but never treated | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN) | Total
Number analyzed (Participants) | 24 | 12 | 52 | 52 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 12 | 50 | 46 | 130
  >=65 years | 2 | 0 | 2 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11.9) | 40 (11.2) | 43 (12.1) | 45 (13.3) | 43 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 10 | 9 | 22
  Male | 22 | 11 | 42 | 43 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 13 | 17 | 41
  Not Hispanic or Latino | 17 | 8 | 39 | 35 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 6 | 25 | 27 | 68
  Black or African American | 13 | 5 | 21 | 16 | 55
  Other or More Than One Race | 1 | 0 | 3 | 5 | 9
  Asian | 0 | 1 | 2 | 1 | 4
  American Indian or Alaska Native | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 12 | 52 | 52 | 140

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 24 as Determined by the US Food and Drug Administration (FDA)-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with the applicable study drug discontinuation status. Week 24 window was between Day 148 and 189 (inclusive). Percentages were rounded off.
Time Frame: Week 24
Population: The Full Analysis Set included all randomized participants who took at least 1 dose of study drug. As none of the participants reached Week 24 timepoint in Cohort 1, data for Cohort 1 were not available for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 52 | 52
percentage of participants |  |  | 1.9 | 0

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 12 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 12 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with the applicable study drug discontinuation status. Week 12 window was between Day 71 and 105 (inclusive). Percentages were rounded off.
Time Frame: Week 12
Population: The participants in the Full Analysis Set were analyzed. As none of the participants were on-treatment in Cohort 1 at Week 12 (required for the analysis of HIV RNA levels using US FDA-defined Snapshot Algorithm), this outcome measure for Cohort 1 could not be analyzed using US FDA-defined Snapshot Algorithm.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 52 | 52
percentage of participants |  |  | 1.9 | 0

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with the applicable study drug discontinuation status. Week 48 window was between Day 316 and 378 (inclusive). Percentages were rounded off.
Time Frame: Week 48
Population: The participants in the Full Analysis Set were analyzed. As none of the participants reached Week 48 timepoint in Cohort 1, data for Cohort 1 were not available for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 52 | 52
percentage of participants |  |  | 0 | 0

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 12 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 12 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with the applicable study drug discontinuation status. Week 12 window was between Day 71 and 105 (inclusive). Percentages were rounded off.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 52 | 52
percentage of participants |  |  | 98.1 [89.7 to 100] | 96.2 [86.8 to 99.5]
Statistical Analysis 1: Comparison: Cohort 2- Group 1 (ISL+LEN) vs Cohort2- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; Difference in percentage = 1.9, 95% CI 2-sided [-6.8 to 11.6] — The difference in percentages between treatment groups and their 95% CI were calculated based on unconditional exact method using 2 inverted 1-sided tests

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with the applicable study drug discontinuation status. Week 24 window was between Day 148 and 189 (inclusive). Percentages were rounded off.
Time Frame: Week 24
Population: The participants in the Full Analysis Set were analyzed. As none of the participants reached Week 24 timepoint in Cohort 1, data for Cohort 1 were not available for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 52 | 52
percentage of participants |  |  | 94.2 [84.1 to 98.8] | 96.2 [86.8 to 99.5]
Statistical Analysis 1: Comparison: Cohort 2- Group 1 (ISL+LEN) vs Cohort2- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; Difference in percentage = -1.9, 95% CI 2-sided [-12.4 to 8.6] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the US FDA-defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with the applicable study drug discontinuation status. Week 48 window was between Day 316 and 378 (inclusive). Percentages were rounded off.
Time Frame: Week 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 52 | 52
percentage of participants |  |  | 96.2 [86.8 to 99.5] | 94.2 [84.1 to 98.8]
Statistical Analysis 1: Comparison: Cohort 2- Group 1 (ISL+LEN) vs Cohort2- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; Difference in percentage = 1.9, 95% CI 2-sided [-8.6 to 12.4] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline in Clusters of Differentiation 4 (CD4)+ Cell Count at Week 12
Time Frame: Baseline and Week 12
Population: The participants from the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 24 | 12 | 52 | 52
cells/µL
  Baseline | 721 (265.0) | 659 (304.8) | 755 (223.6) | 818 (271.3)
  Change at Week 12: number analyzed (Participants) | 19 | 7 | 52 | 50
  Change at Week 12 | -50 (183.0) | 18 (142.3) | -23 (185.6) | -49 (180.0)
Statistical Analysis 1: Comparison: Cohort 1- Group 1 (ISL+LEN) vs Cohort 1- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; p = 0.3859, ANOVA; difference in least squares means = -68, 95% CI 2-sided [-226 to 91] — P-value, difference in least squares means (Diff in LSM), and its 95% confidence interval (CI) were from ANOVA model with treatment group as a fixed effect in the model
Statistical Analysis 2: Comparison: Cohort 2- Group 1 (ISL+LEN) vs Cohort2- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; p = 0.7085, ANCOVA; difference in least squares means = 13, 95% CI 2-sided [-56 to 82] — P-value, difference in least squares means (Diff in LSM), and its 95% CI were from ANCOVA model with baseline value as a covariate and treatment as a fixed effect in the model

8. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline and Week 24
Population: The participants in the Safety Analysis Set with available data were analyzed. As none of the participants reached Week 24 timepoint in Cohort 1, data for Cohort 1 were not available for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 50 | 50
cells/µL |  |  | -4 (182.1) | -57 (204.2)
Statistical Analysis 1: Comparison: Cohort 2- Group 1 (ISL+LEN) vs Cohort2- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; p = 0.3477, ANCOVA; difference in least squares means = 33, 95% CI 2-sided [-37 to 103] — [estimate comment as in outcome 7, analysis 2]

9. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline and Week 48
Population: The participants in the Safety Analysis Set with available data were analyzed. As none of the participants reached Week 48 timepoint in Cohort 1, data for Cohort 1 were not available for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
Number analyzed (Participants) | 0 | 0 | 50 | 49
cells/µL |  |  | -12 (214.7) | -29 (186.1)
Statistical Analysis 1: Comparison: Cohort 2- Group 1 (ISL+LEN) vs Cohort2- Group 2 (B/F/TAF to ISL+LEN); Test type: Other; p = 0.8849, ANCOVA; difference in least squares means = -5, 95% CI 2-sided [-76 to 66] — [estimate comment as in outcome 7, analysis 2]

10. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation
Description: TEAEs were defined as 1 or both of any AEs leading to premature discontinuation of study drug, or any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug. Percentages were rounded off.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Secondary Outcome: Cohort 1: Plasma Concentrations for ISL
Time Frame: Anytime postdose at Week 4
Population: The Pharmacokinetic (PK) Analysis Set for Cohort 1 included all randomized participants who took at least 1 dose of study drug and have at least 1 nonmissing concentration value reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1- Group 1 (ISL+LEN)
Number analyzed (Participants) | 23
ng/mL | 42.1 (49.6)

12. Secondary Outcome: Cohort 2: Pharmacokinetic (PK) Parameter: Cmax of Islatravir (ISL)
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Anytime post dose on Day 1 and at either Week 12 or Week 18
Population: The Pharmacokinetic (PK) Substudy Analysis Set for Cohort 2 included all randomized participants who received at least 1 dose of the study drug, participated in the PK substudy, and had at least 1 nonmissing postdose concentration with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 14
ng/mL
  Day 1: number analyzed (Participants) | 13
  Day 1 | 19.6 (6.55)
  Week 12 or Week 18 | 18.7 (7.6)

13. Secondary Outcome: Cohort 2: PK Parameter: Tmax of ISL
Description: Tmax was defined as the time (observed time point) of Cmax.
Time Frame: Anytime post dose on Day 1 and at either Week 12 or Week 18
Population: The participants in the Pharmacokinetic Substudy Analysis Set for Cohort 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 14
hours
  Day 1: number analyzed (Participants) | 13
  Day 1 | 1.12 (1.03)
  Week 12 or Week 18 | 0.793 (0.423)

14. Secondary Outcome: Cohort 2: PK Parameter: Ctau of ISL
Description: Ctau was defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Anytime post dose at either Week 12 or Week 18
Population: The participants in the Pharmacokinetic Substudy Analysis Set for Cohort 2 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 14
ng/mL | 0.169 (0.0940)

15. Secondary Outcome: Cohort 2: PK Parameter: AUCtau of ISL
Description: AUCtau was defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Anytime post dose at either Week 12 or Week 18
Population: The participants in the Pharmacokinetic Substudy Analysis Set for Cohort 2 were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 14
h*ng/mL | 132 (98.1)

16. Secondary Outcome: Plasma Concentrations for LEN
Time Frame: Anytime postdose at Week 4
Population: The participants in the Pharmacokinetic Analysis Set for Cohort 1 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1- Group 1 (ISL+LEN)
Number analyzed (Participants) | 24
ng/mL | 62.0 (43.9)

17. Secondary Outcome: Cohort 2: Pharmacokinetic (PK) Parameter: Cmax of LEN
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Anytime post dose on Day 1, Day 2 and at either Week 12 or 18
Population: The participants in Pharmacokinetic Substudy Analysis Set for Cohort 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 14
ng/mL
  Day 1: number analyzed (Participants) | 13
  Day 1 | 46.4 (29.0)
  Day 2: number analyzed (Participants) | 13
  Day 2 | 183 (189)
  Week 12 or Week 18 | 97.4 (73.2)

18. Secondary Outcome: Cohort 2: PK Parameter: Tmax of LEN
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Anytime post dose on Day 1, Day 2 and at either Week 12 or Week 18
Population: The participants in the Pharmacokinetic Substudy Analysis Set for Cohort 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 14
hours
  Day 1: number analyzed (Participants) | 13
  Day 1 | 11.4 (8.96)
  Day 2: number analyzed (Participants) | 13
  Day 2 | 6.61 (1.47)
  Week 12 or Week 18 | 5.43 (1.63)

19. Secondary Outcome: Cohort 2: PK Parameter: Ctau of LEN
Description: Ctau was defined as the observed drug concentration at the end of the dosing interval.
Time Frame: Anytime post dose at either Week 12 or Week 18
Population: The participants in the Pharmacokinetic Substudy Analysis Set for Cohort 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 12
ng/mL | 36.6 (22.5)

20. Secondary Outcome: Cohort 2: PK Parameter: AUCtau of LEN
Description: as for outcome 15
Time Frame: Anytime post dose at either Week 12 or Week 18
Population: The participants in the Pharmacokinetic Substudy Analysis Set for Cohort 2 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 2- Group 1 (ISL+LEN)
Number analyzed (Participants) | 12
h*ng/mL | 10000 (7440)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Cohort 1: Up to Week 12; Cohort 2: Up to Week 74.6. Adverse Events: Cohort 1: Up to Week 12; Cohort 2: Up to Week 48
Description: All-cause mortality: All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse events: Safety Analysis Set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Cohort 1- Group 1 (ISL+LEN) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) | Cohort 2- Group 1 (ISL+LEN) | Cohort2- Group 2 (B/F/TAF to ISL+LEN)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12 | 3/52 | 0/52
Other Adverse Events (participants affected / at risk) | 11/24 | 7/12 | 27/52 | 29/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1- Group 1 (ISL+LEN) (N=24) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) (N=12) | Cohort 2- Group 1 (ISL+LEN) (N=52) | Cohort2- Group 2 (B/F/TAF to ISL+LEN) (N=52)
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1- Group 1 (ISL+LEN) (N=24) | Cohort 1- Group 2 (B/F/TAF to ISL+LEN) (N=12) | Cohort 2- Group 1 (ISL+LEN) (N=52) | Cohort2- Group 2 (B/F/TAF to ISL+LEN) (N=52)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 6 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 0 | 3 | 1
Fatigue (General disorders and administration site conditions) | 0 | 0 | 4 | 2
Anal chlamydia infection (Infections and infestations) | 0 | 0 | 3 | 2
Covid-19 (Infections and infestations) | 7 | 2 | 6 | 6
Folliculitis (Infections and infestations) | 1 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 7 | 7
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 3
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (3):
  • Study Protocol: Protocol Amendment 6 (2025-12-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT05052996/Prot_002.pdf
  • Study Protocol: Protocol Amendment 5 (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT05052996/Prot_003.pdf
  • Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT05052996/SAP_001.pdf